CLINICAL TRIAL: NCT05600582
Title: Phase 1 Study of CodaLytic, an Intratumoral Influenza-based Oncolytic Virus, in Patients With Metastatic or Otherwise Inoperable Breast Cancer
Brief Title: A Study of CodaLytic, an Intratumoral Oncolytic Virus, in Patients With Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to funding decision by the sponsor
Sponsor: Codagenix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CDX-ONC-101
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
Keywords: Oncolytic Virotherapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Study participants eligible to participate will be enrolled in each of 4 escalating-dose cohorts and administered intratumoral CodaLytic in the injected lesion during the dosing period as follows: Three (3) doses 4 weeks apart at the low dose, five (5) doses 2 weeks apart at the low dose, three (3) doses 4 weeks apart at the high dose and five (5) doses 2 weeks apart at the high dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 10e7 PFU dose 3 injections (Experimental): 10e7 PFU CodaLytic administered intratumorally once every 4 weeks (3 doses total)
  Interventions: Biological: CodaLytic
- 10e7 PFU dose 5 injections (Experimental): 10e7 PFU CodaLytic administered intratumorally once every 2 weeks (5 doses total)
  Interventions: Biological: CodaLytic
- 10e8 PFU dose 3 injections (Experimental): 10e7 PFU CodaLytic administered intratumorally once every 4 weeks (3 doses total)
  Interventions: Biological: CodaLytic
- 10e8 PFU dose 5 injections (Experimental): 10e8 PFU CodaLytic administered intratumorally once every 2 weeks (5 doses total)
  Interventions: Biological: CodaLytic

INTERVENTIONS:
Biological: CodaLytic — CodaLytic is a virotherapeutic product based on the wild-type influenza strain A/California/07/2009

SUMMARY:
The goal of this phase 1 open label clinical trial is to evaluate the safety and preliminary efficacy of CodaLytic, an intratumorally-administered oncolytic virus, in patients with metastatic or otherwise inoperable breast cancer.

The main questions it aims to answer are:

* How safe is CodaLytic when administered in escalating dosing groups into targeted lesions?
* What is the impact of CodaLytic on lesion response and disease progression?

Eligible participants will be enrolled into four (4) escalating dose groups and treated with Codalytic through injection into a selected lesion(s) over twelve (12) weeks and then followed for up to one (1) year after the first dose. A safety committee will review the safety profile of each dosing group before the next dose-escalation.

Study procedures will include physical examinations, injection site assessments, biopsies, imaging, and collection of blood/urine to assess safety, the body's immune response, and efficacy.

DETAILED DESCRIPTION:
This study is a Phase 1, open-label, 3+3 dose-escalation, clinical trial to evaluate the safety and preliminary efficacy of CodaLytic in patients with metastatic or otherwise inoperable breast cancer.

After providing informed consent, screened participants will undergo baseline safety assessment and imaging. The Investigator will select an accessible lesion for intratumoral injection of CodaLytic (the injected lesion), and a core needle biopsy sample of this lesion will be obtained for eligible participants to be dosed. The Investigator will also select additional lesions for imaging (target lesions); these target lesions will not be injected or biopsied. If possible, another accessible lesion that is not a target lesion will be selected for biopsy to assess abscopal effect.

Three (3) eligible participants who meet all study inclusion and no exclusion criteria will be enrolled in each of four (4) escalating-dose cohorts and administered intratumoral CodaLytic. Up to 3 additional participants per cohort may be enrolled. During the dosing period, participants will be assessed for adverse events, serious adverse events, and dose-limiting toxicities. A safety review committee will review the safety data through Day 28 for the participants in Cohort 1 before participants are enrolled in Cohorts 2 and 3 and safety data through Day 28 for the participants in Cohorts 2 and 3 before participants are enrolled in Cohort 4. The safety review committee will also meet on an ad hoc basis to review any unexpected safety concerns.

Enrolled participants will be followed for adverse events, serious adverse events, dose-limiting toxicities to assess safety of CodaLytic administration. Biopsy samples of the injected lesion and, if possible, from a noninjected, nontarget lesion will be collected at Week 5. At the end of treatment, imaging will be performed for staging by Response Evaluation Criteria in Solid Tumours (RECIST) 1.1, and biopsy samples will be collected. Repeat disease assessment will be performed 4 to 8 weeks after the Month 3/EOT visit if complete response (CR) or partial response (PR) is observed at that visit or if progressive disease (PD) is seen at that visit and the participant has not begun additional cancer treatment. After the treatment period, participants may enroll in other studies or be managed with other treatment modalities as indicated, but follow-up assessments of Investigator-assessed tumor response and anticancer treatments will be recorded at Months 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Women or men with metastatic or inoperable, histologically confirmed breast cancer
* Has no alternative treatment of proven benefit available or has refused treatment
* Expected survival ≥ 3 months
* At least 2 measurable lesions according to RECIST 1.1, without contraindication for repeated injections and core needle biopsies
* Adequate organ function
* Eastern Cooperative Oncology Group performance status of 0 to 2
* Negative pregnancy test, if female
* Agreement to practice a highly effective method of contraception
* Agreement to no sperm donation through 28 days, if male
* Willing to provide consent to perform study procedures

Exclusion Criteria:

* Pregnant or lactating women
* Anticancer therapy within 3 weeks of dosing
* Known active central nervous system metastases (with some exceptions)
* Presence of a concurrent malignancy for which the natural history or treatment has the potential to interfere with the safety or efficacy assessment of the Investigational Product
* Uncontrolled or severe cardiovascular disease
* Immunodeficiency or use of therapies expected to impair the immune response within thirty (30) days of enrollment or during dosing.
* Ongoing toxicity > Grade 1 from prior treatment except those which are stable
* History of severe reaction (ie, anaphylaxis) to vaccination or immunotherapy
* Planned radiation to lesions targeted for assessment/injection within 60 days before first dose or any planned radiation during dosing period
* Any condition or occupational or other responsibility that in the judgment of the Investigator would interfere with or serve as a contraindication to protocol adherence, assessment of safety, or a participant's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
To assess the Serious Adverse events (SAEs) of CodaLytic administered by intratumoral injection | Dosing Period approximately 3 months from first dose
  To assess the frequency of Serious Adverse events (SAEs) of CodaLytic administered by intratumoral injection at 2-weekly or 4-weekly intervals at doses of 10e7 and 10e8 plaque-forming units (PFU)/mL
To assess the Adverse events (AEs) of CodaLytic administered by intratumoral injection | Dosing Period approximately 3 months from first dose
  To assess the frequency of Adverse events (AEs) of CodaLytic administered by intratumoral injection at 2-weekly or 4-weekly intervals at doses of 10e7 and 10e8 plaque-forming units (PFU)/mL
To assess the Dose-limiting toxicities (DLTs) of CodaLytic administered by intratumoral injection | Dosing Period approximately 3 months from first dose
  To assess the frequency of Dose-limiting toxicities (DLTs) of CodaLytic administered by intratumoral injection at 2-weekly or 4-weekly intervals at doses of 10e7 and 10e8 plaque-forming units (PFU)/mL

SECONDARY OUTCOMES:
CodaLytic administration impact on tumor response and disease progression: Overall response rate (ORR) | 3 months, 6 months, and 12 months from treatment
  To assess the Overall response rate (ORR) for CodaLytic intratumoral administration as a measurement of tumor response and disease progression
CodaLytic administration impact on tumor response and disease progression: Duration of response (DoR) | 3 months, 6 months, and 12 months from treatment
  To assess the Duration of response (DoR) for CodaLytic intratumoral administration as a measurement of tumor response and disease progression
CodaLytic administration impact on tumor response and disease progression: Disease control rate (DCR) | 3 months, 6 months, and 12 months from treatment
  To assess the Disease control rate (DCR) for CodaLytic intratumoral administration as a measurement of tumor response and disease progression
CodaLytic administration impact on tumor response and disease progression: Progression-free survival (PFS) | 6 months, and 12 months from treatment
  To assess the Progression-free survival (PFS) for CodaLytic intratumoral administration as a measurement of tumor response and disease progression

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Gabrail Cancer Center, Canton, Ohio

IPD SHARING:
Plan to Share IPD: No